CLINICAL TRIAL: NCT06700486
Title: Clinical and Radiographic Assessment of the Socket Shield Technique Accompanied by Sticky Bone Around the Immediate Implant
Brief Title: Assessment of the Socket Shield Technique Accompanied by Sticky Bone Around the Immediate Implant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reham Qabeel (Other)
Responsible Party: Sponsor-Investigator, Reham Qabeel, Assistant lecturer, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: P-ME-22-02
Record Dates: First submitted 2022-07-31; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Immediate Implant
Keywords: socket shield; sticky bone
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comparator arm (Active Comparator): Immediate implant and sticky bone
  Interventions: Procedure: SOCKET SHIELD
- interventional arm (Other): Socket shield
  Interventions: Procedure: Immediate implant and sticky bone

INTERVENTIONS:
Procedure: SOCKET SHIELD — in implant dentistry
  Arms: comparator arm
Procedure: Immediate implant and sticky bone — in implant dentistry
  Arms: interventional arm

SUMMARY:
challenge of the implant of esthetic zone with buccal plate of bone width less than 2mm become available by the using of socket shield technique used with the immediate implant this technique provide improvement of the width of buccal plate of bone which improve esthetic outcome bot the jumping gape still a questionable area between the shield and the implant which required to be filled with biological filling to improve osteointegration and stability of the implant such as sticky bone ,bone mixed with injectable PRF , PRF also has antibacterial ,anti-inflammatory effect and regenerative effect which could help.

DETAILED DESCRIPTION:
Biological mechanisms involved in the healing of the periodontal tissues after tooth extraction can cause the loss of the periodontal ligament and its vascular support. The physiological process can lead to esthetic problems that are difficult to resolve by methods of restoration that are able to preserve the emergence profile, especially in the anterior region . Therefore, preserving and maintaining the bone anatomy and soft tissue architecture in the anterior region is essential for maintaining esthetics restorations .

Teeth extractions basis volumetric changes characterized by alveolar bone resorption, specifically the buccal plate of bone, with a consequential associated soft tissue retraction . Several studies proved that buccal dimension of the alveolar ridge undergoes horizontal bone resorption of about 56% and a resorption of the palatal /lingual bone of 30% through the interval four-month prior extraction of the tooth. Correspondingly . detected overall horizontal dimension resorption of the alveolar ridge subsequent the extraction, and the buccal wall reduction of the alveolar ridge is more obvious than lingual wall .

Immediate placement of implant does not totally overcome the resorption of the alveolar bone and recession of the soft tissue in esthetic region following teeth extractions. Loss of alveolar bone prior extraction consider as irreversible process concerning both vertical and horizontal resorption. Moreover, the alveolar bone resorption is more distinct on the buccal wall than on the lingual wall of the extraction socket.

The ridge dimension is reduced when implants are placed immediately without subsequent directed bone regeneration treatments. When compared to spontaneous healing, it appears to be ineffective at around half of the initial bone width in horizontal dimension . By using a grafting substance and combining instantaneous implant insertion with a guided bone-regeneration process, less horizontal bone resorption can be expected .

Several augmentation techniques are used in the surgical field to create sufficient bone volume. Grafting techniques for particulate bone augmentation include autograft, allograft, xenograft, and alloplast. Autograft is the gold standard in bone augmentation, but it has drawbacks such as second surgical-site morbidity and insufficient bone volume. Secondary infections are a disadvantage of allografts and xenografts Since 2010, a novel method of producing growth factor-enriched bone graft matrix (also known as sticky bone) with autologous fibrin glue has been demonstrated. Sticky bone stabilizes the bone graft in the defect, accelerating tissue healing and minimizing bone loss during the healing period. It is moldable and adaptable to a variety of bony defects, preventing micro and macro movement of the grafted bone. As a result, the volume of the augmentation is maintained during the healing process, and the need of titanium mesh and bone block is reduced .

In contrast to PRP or PRGF, the fibrin network entraps platelets and leukocytes to release growth factors, speeding up soft tissue regeneration and bone regeneration. Furthermore, unlike PRP or PRGF, no biochemical additives are required to make sticky bone, and fibrin interconnection reduces soft tissue ingrowth into the sticky bone graft .

Studies revealed that the presence of vascular supply from the periodontal ligament was a major factor in the preservation of alveolar bone and soft tissues, the idea of leaving the leftover root section on the labial plate was advocated. This procedure is known as "socket shield technology" in which the root fragment acts as a shield to protect the buccal bone from resorption

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients having at least single tooth into esthetic zone indicated for extraction and immediate implant placement.

2. patient with adequate oral hygiene and systemically free. 3.patients' age ranging from 20-60 years. 4. Free from any systemic disease according to Cornell Medical Index

Exclusion Criteria:

* 1. Presence of para-functional habits such as bruxism, clenching, excessive gum chewing, lip or fingernail biting.

  2. Chronic smokers or formal smoker. 3.Insulin dependent diabetes 4.Thyroid disease 5.Clinical diagnosis of Alzheimer's Disease 6. patients receiving chemotherapy or radiotherapy, alcohol or drug abuse 7. Pregnancy and lactation.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue thickness | 6 months
  measured with mm
Marginal bone loss | 9 months
  measured with mm

SECONDARY OUTCOMES:
Buccal bone width | 6 and 9 months
  width measured with mm
Buccal bone length | 6 and 9 months
  length measured with mm
Bone density | 6 and 9 months
  Bone density measured with Hounsfield index

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Abdel Hady Ali Kabeel, Cairo, Egypt